CLINICAL TRIAL: NCT02182583
Title: A Phase III Study of Ba253BINEB in Patients With COPD - Double-blind, Randomised, Double Dummy, Multiple Dose Study in Comparison With MDI
Brief Title: Ba253BINEB Compared to Ba253MDI (Metered Dose Inhaler) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54.560
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Ba253BINEB (Experimental)
  Interventions: Drug: Ba253BINEB
- Ba253MDI (Active Comparator)
  Interventions: Drug: Ba253MDI

INTERVENTIONS:
Drug: Ba253MDI
  Other Names: Tersigan® aerosol
  Arms: Ba253MDI
Drug: Ba253BINEB
  Arms: Ba253BINEB

SUMMARY:
The objective of this study is to investigate the efficacy and safety of Ba253BINEB during the continuous 4 weeks administration to the patients with COPD using Ba253MDI (Tersigan® aerosol) as the comparator drug.

ELIGIBILITY:
Inclusion Criteria:

The patients with COPD (chronic bronchitis, emphysema) and who satisfy the following criteria

1. Patients whose symptoms are stable and have at least 4 symptomatic days a week
2. Patients with FEV1.0/FVC of <= 70% in the screening test
3. Patients aged >= 40 years or older
4. Patients must be able to inhale the study drug via BINEB and MDI
5. Patients must be able to understand the patient information form

Exclusion Criteria:

Those who correspond to the following shall be excluded from the subjects of study.

1. Patients complicated with bronchial asthma, making the assessment of drug efficacy against COPD difficult
2. Patients who are constantly administered oral steroid
3. Patients with glaucoma
4. Patients who have prostatic hypertrophy
5. Patients with hypersensitivity to anticholinergic drugs or Beta2 agonists.
6. Patients with serious hepatic disease, kidney disease or heart disorder and who are judged by the investigator as inappropriate as the subjects of study
7. Women who are pregnant or who may become pregnant, or nursing women
8. Patients who are judged by the investigator as inappropriate as the subjects of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 1998-10; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Change in COPD daily symptom scores | Baseline and up to 4 weeks after first drug administration

SECONDARY OUTCOMES:
Change from baseline in times of cough | Baseline, up to 4 weeks after first drug administration
Change from baseline in peak expiratory flow rate (PEFR) | Baseline, up to 4 weeks after first drug administration
Number of Patients with Adverse Events | Up to 4 weeks
Number of patients with significant changes in vital sings (blood pressure, pulse rate) | Baseline, week 4
Number of patients with abnormal changes in electrocardiogram (ECG) | Baseline, week 4
Number of patients with abnormal changes in laboratory values | Baseline, week 4
Physician's global evaluation | 4 weeks after first drug administration
Patient's impression | 4 weeks after first drug administration
Change from baseline in times and volume of sputum | Baseline, up to 4 weeks after first drug administration
Change from baseline in transition of nocturnal sleep | Baseline, up to 4 weeks after first drug administration
Change from baseline in FEV1 (Forced expiratory volume in one second) | Baseline, week 4
Change from baseline in FVC (Forced vital capacity) | Baseline, week 4